CLINICAL TRIAL: NCT05717101
Title: Contrast-Enhanced Harmonic Endoscopic Ultrasound Imaging - a Patient Registry
Brief Title: Patient Registry in Patients Undergoing Contrast-Enhanced Harmonic Endoscopic Ultrasound Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-008737; NCI-2022-11067 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-01-12; First posted 2023-02-08 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2023-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical records): Patients who have undergo contrast-enhanced harmonic endoscopic ultrasound imaging have their medical records reviewed.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study creates a patient registry of patients undergoing contrast-enhances-harmonic endoscopic ultrasound imaging. In order to improve what doctors see on the ultrasound exam, sometimes intravenous contrast can be used to better emphasize the blood flow in a particular organ or lesion. Creating a local database that can be used as a patients registry may help doctors keep track of all patients that undergo contrast-enhanced endoscopic ultrasound procedures and also to monitor for possible procedure adverse events.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the findings and outcomes of patient undergoing contrast-enhanced harmonic endoscopic ultrasound (CE-EUS) imaging.

OUTLINE: This is an observational study.

Patients who have undergo contrast-enhanced harmonic endoscopic ultrasound imaging have their medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years to 99 years old who were undergo CE-EUS are eligible for study inclusion
* Based on clinical judgement of the advanced endoscopist will include those who present with lesions where increased microvasculature and perfusion visualization with contrast-enhanced harmonic endoscopic ultrasound imaging would be of beneficial for lesion characterization
* Clinical medical stability to undergo sedation for endoscopy and provide informed consent

Exclusion Criteria:

* Medical condition that preclude the patient from having an endoscopic procedure
* Patients who cannot provide adequate research authorization
* Patients with known allergies to ultrasound contrast agents
* Patient who did not receive contrast during endoscopic ultrasound (EUS) exams

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo contrast-enhanced harmonic endoscopic ultrasound imaging in the gastroenterology department at Mayo Clinic Jacksonville, Florida
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Analyse continuous variable outcomes of patient undergoing contrast-enhanced harmonic endoscopic ultrasound imaging using medical record review and T-tests or Mann-Whitney U test. | Up to 5 years
  Descriptive statistical analysis will be carried out at routine intervals for database analysis. Two-sided P values less than 0.05 will be considered statistically significant. For descriptive analyses, continuous variables will be reported as a mean +/- standard deviation or median (interquartile range) and compared based on either T-tests or Mann-Whitney U test.
Analyse categorical variable outcomes of patient undergoing contrast-enhanced harmonic endoscopic ultrasound imaging using medical record review and chi-square test or Fisher's exact test. | Up to 5 years
  Descriptive statistical analysis will be carried out at routine intervals for database analysis. Two-sided P values less than 0.05 will be considered statistically significant. Categorical variables will be reported as frequencies with percentages and compared using the chi-square test or Fisher's exact test.
Analyse multivariables of patient undergoing contrast-enhanced harmonic endoscopic ultrasound imaging using medical record review and logistic regression or linear regression analyses depending on the outcome. | Up to 5 years
  Descriptive statistical analysis will be carried out at routine intervals for database analysis. Two-sided P values less than 0.05 will be considered statistically significant. Multivariable analyses will be performed using logistic regression or linear regression analyses depending on the outcome, i.e. dichotomous or continuous respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States